CLINICAL TRIAL: NCT07032649
Title: Double-Blind, Placebo-Controlled Clinical Trial Evaluating Benzoyl Peroxide for Preventing Recurrence of HSV-1 Outbreaks With Rescue Crossover Option
Brief Title: Evaluating Benzoyl Peroxide for Preventing Recurrence of HSV-1 Outbreaks With Rescue Crossover Option
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Greg Bew (Industry)
Responsible Party: Sponsor-Investigator, Greg Bew, Clinical Research Coordinator, Erroll McCoy
Organization: Erroll McCoy (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EM202501
Record Dates: First submitted 2025-06-16; First posted 2025-06-24 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: HSV
Keywords: HSV; HSV-1; HSV suppression; Herpes
MeSH Terms: conditions — Herpes Simplex | interventions — Benzoyl Peroxide; Receptors, Catecholamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Treatment (Experimental): 10% Benzoyl Peroxide topically applied
  Interventions: Drug: Benzoyl Peroxide 10% Bar
- Placebo Arm (Placebo Comparator): Placebo applied topically
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Benzoyl Peroxide 10% Bar — Active ingredient for drug included. Blind identification by package number
  Arms: Active Treatment
Other: Placebo — Placebo that looks like active treatment, blinded but available to ID via package number
  Arms: Placebo Arm

SUMMARY:
Here's a clear, concise, and accurate **brief summary** suitable for your ClinicalTrials.gov PRS submission:

* Brief Summary:

This randomized, double-blind, placebo-controlled clinical trial evaluates the effectiveness of topical Benzoyl Peroxide (10%) in preventing recurrent oral lesions caused by Herpes Simplex Virus Type 1 (HSV-1). Participants who experience frequent HSV-1 outbreaks will be randomly assigned to either Benzoyl Peroxide or placebo treatment. The trial will be conducted via telehealth visits, with treatment provided remotely. The primary objective is to determine whether Benzoyl Peroxide significantly delays or prevents HSV-1 lesion recurrence compared to placebo. Secondary outcomes include evaluating recurrence frequency, lesion severity, healing duration, and participant satisfaction. The trial also incorporates a rescue crossover step, allowing placebo-group participants who experience recurrence to receive active treatment. Results from this pilot study will inform the potential use of Benzoyl Peroxide as a novel, accessible topical treatment option for recurrent HSV-1 outbreaks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled clinical trial investigating the effectiveness of topical Benzoyl Peroxide 10% cream in preventing the recurrence of oral lesions (cold sores) caused by Herpes Simplex Virus Type 1 (HSV-1). The study is designed as a small-scale, pilot clinical trial conducted entirely via telehealth appointments, with treatment and placebo creams shipped directly to enrolled participants.

Participants aged 18-65 with a documented history of at least two HSV-1 outbreaks per year will be enrolled and randomized into two groups:

* **Active Treatment Group**: Receives topical Benzoyl Peroxide 10% cream.
* **Placebo Group**: Receives an identical topical cream formulation without the active ingredient.

All participants will be instructed to apply the assigned topical cream twice daily (morning and evening) at the onset of HSV-1 symptoms for a minimum of five days, continuing until lesions fully resolve or up to a maximum of 14 days.

The primary objective of this clinical trial is to evaluate the efficacy of Benzoyl Peroxide 10% cream in extending the time until the recurrence of HSV-1 outbreaks within a 6-month follow-up period compared to placebo.

Secondary outcomes include:

* Evaluating the frequency of HSV-1 recurrences within 6 months.
* Measuring the severity and duration of lesions and associated pain.
* Determining participant satisfaction and overall treatment acceptability.
* Assessing the effect of lesion anatomical location on recurrence patterns.

A unique aspect of this trial is the inclusion of a **rescue crossover procedure**, where participants initially randomized to placebo who experience a confirmed recurrence at the previously treated site will be provided Benzoyl Peroxide 10% cream, ensuring ethical access to potentially effective treatment.

To ensure unbiased trial conduct and data integrity, oversight measures have been implemented, including:

* Independent Clinical Research Coordinator (with no financial interest) responsible for auditing data accuracy, protocol adherence, and regulatory compliance.
* Supervising Physician (with no financial interest) providing clinical oversight and quality assurance of trial activities conducted by the Principal Investigator.

Results from this trial aim to inform the potential efficacy and safety profile of Benzoyl Peroxide as a topical therapy for HSV-1 recurrence prevention, potentially supporting future FDA regulatory submissions or larger-scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-65 years, inclusive.

Documented history of at least two HSV-1 outbreaks per year.

Ability and willingness to participate fully via telehealth (including video visits).

Must provide informed consent to participate in the trial.

Ability to comply with the trial protocol, including symptom reporting, topical cream application, and follow-up telehealth appointments.

Exclusion Criteria:

Currently pregnant or breastfeeding, or plans to become pregnant during the study period.

Known allergy or sensitivity to benzoyl peroxide or similar topical agents.

Current participation in another clinical trial involving topical treatments.

Medical conditions or skin conditions that could significantly interfere with topical treatment application or safety assessment.

Inability to effectively participate in telehealth visits or use video-based symptom verification.

Participants who, in the opinion of the investigator, are unlikely to comply fully with trial requirements or complete the 6-month follow-up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Time to First Recurrence of HSV-1 Outbreaks Within 6 Months | 6 months
  The primary outcome measure is the duration of time (measured in days) from initial treatment application until the participant experiences the first confirmed recurrence of an HSV-1 lesion. Recurrence is confirmed through telehealth video consultation and visual verification by the study team. The maximum observation period for each participant is 6 months following initial treatment. The effectiveness of topical Benzoyl Peroxide (10%) versus placebo in prolonging recurrence-free intervals will be evaluated using Kaplan-Meier analysis.

CONTACTS AND LOCATIONS:
Overall Officials: David Dinn, DMSc, Principal Investigator — Erroll McCoy
Locations (1):
- Zoom Health, Telehealth Only, Evans, Georgia, United States

IPD SHARING:
Plan to Share IPD: No